CLINICAL TRIAL: NCT06847477
Title: SOFA Score with Serum Procalcitonin Versus SOFA Score with Neutrophil/lymphocyte Ratio in Predicting Sepsis and Clinical Outcomes in Intensive Care Unit.
Brief Title: SOFA Score with Serum Procalcitonin Versus SOFA Score with Neutrophil/lymphocyte Ratio in Predicting Sepsis and Clinical Outcomes in I.C.U.
Acronym: SOFA-PROVSNL
Status: Not yet recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU R24/2025
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Sepsis; Critical Illness
Keywords: SOFA score; procalcitonin; neutrophils to lymphocytes ratio
MeSH Terms: conditions — Sepsis; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Critically ill patients presented to Surgical and Trauma intensive care: Critically ill patients who are presented to the Surgical and Trauma intensive care unit will be assessed on admission to ICU by SOFA score, procalcitonin, and neutrophils/lymphocytes ratio.
  then the patients will be followed to measure the length of stay and mortality.

SUMMARY:
Sepsis remains a critical life-threatening and a healthcare challenge worldwide. Sepsis is implicated in a mortality rate that ranges between 25 - 30% in severe cases and 40-70% in septic shock, also, Post sepsis, lower quality of life was observed among survivors, therefore early prediction and a rapid therapeutic decision, are essential to improve patient outcomes.

Different indicators are proposed as predictors but with different sensitivity, specificity, and availability. This study aims to evaluate the efficacy of PCT and SOFA scores versus SOFA and NLR in predicting morbidity and mortality outcomes in sepsis.

DETAILED DESCRIPTION:
Sepsis provokes a dysregulated host response to infection that leads to acute organ dysfunction. The subsequent Septic shock, which includes an underlying circulatory and cellular imbalance increases the mortality. Septic shock manifests as persistent hypotension requiring vasopressors to maintain a mean arterial pressure of 65 mm Hg or higher and a serum lactate level greater than 2 mmol/L (18 mg/dL) in the absence of hypovolemia.

Sequential Organ Failure Assessment score (SOFA) has become extensively used and one of the gold standard tests in assessing the patient's status during intensive care unit (ICU) stay and predicting the clinical outcomes of the patients, however, poor sensitivity of SOFA score is a major limitation that excludes its use as a screening tool for early sepsis, the stage in which treatment is most effective. Blood culture is a well-established diagnostic test for sepsis, however, has limitations e.g. prolonged incubation time and probability of false-negative results.

Procalcitonin (PCL) has been studied as a sepsis biomarker, to help with sepsis diagnosis and to guide the initiation and cessation of antibiotics. Procalcitonin strongly correlates with the extent and severity of bacterial infections, better indicator of illness severity than CRP, and also, provides a quick result compared to blood cultures. Procalcitonin use may be hindered by availability and the cost in a limited resources environment, However, The neutrophil-to-lymphocyte ratio (NLR) is a readily available marker. The neutrophil-to-lymphocyte ratio (NLR) is an indicator of systemic inflammation based on complete blood count values. In general, blood neutrophil count increases with the progress of the inflammatory disease, NLR is more reliable when predicting patient survival than either neutrophil count or lymphocyte count alone.

Endogenous cortisol and catecholamines increase the neutrophil count while simultaneously decreasing the lymphocyte count so it may be major drivers of the NLR. Also, cytokines and other hormones are likely to be involved. So NLR is not solely an indication of infection or inflammation. Any cause of physiologic stress may increase the NLR (e.g. hypovolemic shock). NLR increases rapidly following acute physiologic stress (<6 hours). This prompt response time may make NLR a better reflection of acute stress. Interpretation of NLR level is as follows: A normal NLR is roughly 1-3, An NLR of 6-9 suggests mild stress and Critically ill patients will often have an NLR of ~9 or higher (occasionally reaching values close to 100).

This research will test the predictability of combined SOFA score and procalcitonin versus combined SOFA score and NLR for clinical outcomes such as length of ICU stay and mortality.

ELIGIBILITY:
Inclusion Criteria:

* critically ill patients admitted to ICU for surgical or trauma causes.

Exclusion Criteria:

* Lack of consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients presented to Surgical and Trauma intensive care unit
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Length of ICU stay | from the time of admission to the time of discharge from the ICU or death up to 40 days from ICU admission
  It includes the total number of days spent in the ICU, calculated from the time of admission to the time of discharge from the ICU or death, whichever comes first.
  The unit of measurement is days.

SECONDARY OUTCOMES:
28 days mortality | From the day of admission at the ICU and up to 28 days.
  the occurrence of the event of mortality. It will be followed from the day of admission at the ICU and up to 28 days
Antibiotics used | From ICU admission to discharge from ICU or death which comes first up to 40 days from admission.
  Duration and number of antibiotic usage: measured by the time of the first dose of antibiotics till the time of the last dose administration in the ICU.

IPD SHARING:
Plan to Share IPD: Undecided
May be shared under reasonable request

REFERENCES:
- [Background] Kumar R, Kattimani B, Ojha PR, Khasage UJ. Quick Sequential Organ Failure Assessment Score, Lactate, and Neutrophil-Lymphocyte Ratio Help in Diagnosis and Mortality Prediction during Golden Hour of Sepsis in Emergency Department. J Emerg Trauma Shock. 2023 Oct-Dec;16(4):161-166. doi: 10.4103/jets.jets_37_23. Epub 2023 Oct 24. PMID 38292274
- [Background] Bajic D, Matijasevic J, Andrijevic L, Zaric B, Lalic-Popovic M, Andrijevic I, Todorovic N, Mihajlovic A, Tapavicki B, Ostojic J. Prognostic Role of Monocyte Distribution Width, CRP, Procalcitonin and Lactate as Sepsis Biomarkers in Critically Ill COVID-19 Patients. J Clin Med. 2023 Feb 2;12(3):1197. doi: 10.3390/jcm12031197. PMID 36769843